CLINICAL TRIAL: NCT05682573
Title: Study on Immune Status of Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: Qilu-20230105-pang
Record Dates: First submitted 2023-01-07; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Immunity; Life Quality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml*4 blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid-19 Inpatients: Participant is diagnosed with symptomatic COVID-19 by a positive polymerase chain reaction(PCR) or rapid antigen detection for SARS-CoV-2 and with treatment in hospital
  Interventions: Diagnostic Test: hospitalized patient

INTERVENTIONS:
Diagnostic Test: hospitalized patient — Collect the patient's whole blood for testing

SUMMARY:
This study is a prospective cohort study aimed to clarify the continuous immune state changes of patients with COVID-19. Investigators include the patients admitted to the hospital within one week after the onset of COVID-19. 10ml of patients' blood was collected day 1, day 7, day 14 , and day 20 after the patients admitted to the hospital. The blood inflammatory factors, immune related molecules, and immune cells were detected to determine the changes of patients' immune status. The impact of immune status changes on prognosis and quality of life in later follow-up period was evaluated by various questionnaires and evaluation scales.

DETAILED DESCRIPTION:
After SARS-CoV-2 infection, the patient's immune system is overactivated. While the immune cells release a large number of proinflammatory factors, anti-inflammatory response starts at the same time. Anti-inflammatory factors such as interleukin 4 (IL-4), interleukin 10 (IL-10) and interleukin 37 (IL-37) will be compensated to resist the release of proinflammatory factors and prevent the further development of systemic inflammatory response. However, when the anti-inflammatory factor is excessively released, it will cause compensatory response syndrome, leading to immunosuppression. Whether the level of anti-inflammatory factors continues to rise, and whether it will lead to the persistence of later immunosuppression is unknown. Therefore, this study intends to recruit patients infected with novel coronavirus to enter the hospital within one week of onset, and collect 10ml of patients' blood on the first, seventh, fourteenth and twentieth day after the patients feel the hospital feeling, respectively, to detect the blood inflammatory factors, immune related molecules and immune cells, and determine the changes of patients' immune status. The patients were followed up for 2 and 6 months after arriving at the hospital to conduct self-reported symptom questionnaire, health related quality of life (HRQoL) questionnaire, Hospital Anxiety and Depression Scale (HADS), and other questionnaires and scales to assess the impact of changes in the patient's immunological status on the prognosis and later quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as novel coronavirus infection by PCR or antigen rapid detection for the first time
2. Patients hospitalized within one week after the occurrence of clinical symptoms related to novel coronavirus infection (fever, cough, shortness of breath or dyspnea, fatigue, headache, muscle or body pain, sore throat, nasal congestion or runny nose, chills, nausea, vomiting, diarrhea, mental state changes)
3. Age over 18, gender unlimited

Exclusion Criteria:

1. Patients with immunosuppression, including HIV infection, hematopoietic stem cell transplantation and high-dose immunosuppressant therapy
2. Patients with severe autoimmune diseases
3. Patients receiving chemotherapy or cancer treatment
4. Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant is diagnosed with symptomatic COVID-19 by a positive PCR or rapid antigen detection for SARS-CoV-2 and with treatment in hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-05 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the concentration of inflammatory markers (IL-1β、IL-2、 IL-2R 、IL-4 、 IL-6 、 IL-8、 IL-10 、 interferon-gamma（IFN-γ）、tumour necrosis factor alpha(TNF-α) 、vascular endothelial growth factor（VEGF）, etc.) in peripheral blood. | 1, 7, 14, 20 days after the patient arrives at the hospital
Changes in the concentration of immunosuppression makers(HLA-DR, Programmed Cell Death Ligand 1 （PD-1）, T cell immunoglobulin and mucin domain 3（TIM-3）,etc.) in peripheral blood. | 1, 7, 14, 20 days after the patient arrives at the hospital
Changes in the number of immune cells(Th1/Th2 cell, Treg cell, Myeloid-derived suppressor cells,etc.) in peripheral blood. | 1, 7, 14, 20 days after the patient arrives at the hospital

SECONDARY OUTCOMES:
self-reported symptom | 2，6 months after the patient arrives at the hospital
health related quality of life (HRQoL) questionnaire, | 2，6 months after the patient arrives at the hospital
  There are five dimensions, each with a minimum value of 1 and a maximum value of 3, and the higher score mean a worse outcome
Hospital Anxiety and Depression Scale (HADS) | 2，6 months after the patient arrives at the hospital
  There are two dimensions, each with a minimum value of 0 and a maximum value of 21，and higher score mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No